CLINICAL TRIAL: NCT04822727
Title: A Prospective Physician-Initiated PMCF Study Investigating the Safety and Clinical Performance of the Lokum L-Quest Guidewire, the Lokum Amplatz Guidewire, the Slider Hydrophilic Nitinol Guidewire, the AltoSa-XL PTA Balloon, the AltoSa-XL Gemini Balloon Catheter, the Optimus XL CoCr Stent and the Optimus CVS PTFE Covered XL Stent for the Endovascular Intervention
Brief Title: AndraTec PMCF Study : Investigating the AndraTec Guidewires,PTA Balloons and Stents in Iliac Disease.
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor did not pusue with the study
Sponsor: Dr. Sabrina Overhagen (Other)
Responsible Party: Sponsor-Investigator, Dr. Sabrina Overhagen, Study Director, FCRE (Foundation for Cardiovascular Research and Education)
Organization: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Other Study IDs: FCRE-201016
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Iliac Artery Disease; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 1 or more AndraTec devices (see description for list of devices) — 1 or more AndraTec devices (Lokum L-Quest guidewire, Lokum Amplatz guidewire, Slider Hydrophilic Nitinol Guidewire, AltoSa-XL PTA Balloon, Alto-Sa-XL Gemini Balloon, Optimus-CoCr stent, Optimus-CVS PTFE covered stent)

SUMMARY:
This PMCF study is designed as prospective, multi-center study to collect real-life data.

The rationale of this study is to confirm and support the clinical safety and performance of the aforementioned products in 200 patients who will undergo an endovascular intervention within standard-of-care (SOC) where at least 1 of the following devices from AndraTec were used:

The LOKUM-Quest guidewire, The LOKUM AMPLATZ guidewire, the Slider Hydrophilic Nitinol Guidewire, the AltoSa-XL PTA balloon, the AltoSa-XL GEMINI PTA Balloon, the OPTIMUS CoCr Stent , the OPTIMUS-CVS PTFE-Covered stent.

ELIGIBILITY:
Inclusion Criteria:

- Corresponding to the CE-mark indications/contra-indications and according to the current medical guidelines for minimally invasive peripheral interventions.

Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study (depending on the used device during the procedure) Patient is >18 years old Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study Patient is eligible for treatment with

* the Lokum L-Quest guidewire
* and/or the Lokum Amplatz guidewire
* and/or the Slider Hydrophilic Nitinol Guidewire
* and/or the AltoSa-XL PTA balloon
* and/or the AltoSa-XL Gemini balloon catheter
* and/or the Optimus-XL CoCr Bare Metal Stent
* and/or the Optimus-XL CVS PTFE Covered Stent, as described in the IFU for each device.

Exclusion Criteria:

* Application in coronary, cerebral arteries and central circulatory system
* Known contraindication to peripheral arterial and visceral vasculature treatment - Anatomy or size of vessels that will not allow appropriate usage of the investigational devices, following IFU of the investigational devices.
* Known contraindication and/or allergy to (a component of) an investigational device
* Pregnant women and women with childbearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow-up period.

Device-related exclusion criteria (not applicable for guidewire):

* Known contraindications given in the IFU of Optimus CoCr and Optimus-CVS PTFE- Covered Balloon-Expandable Stent which includes treatment of renal arteries, aneurysms adjacent to site of stent implantation and neurovascular treatment
* Known contraindications given in the IFU of AltoSa-XL-PTA and AltoSa-XL-Gemini Balloon catheter:

  * patients with a contraindication for anti-platelet/anti-coagulant therapy
  * patients with excessive vessel tortuosity
  * dilatation of in-stent restenosis and highly calcified stenosis
  * patients with perforated vessels evidenced by extravasation of contrast media
  * patients with a known hypersensitivity to nylon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease, meeting the in/exclusion criteria and eligible for treatment with the AndraTec devices, according to the IFU of each device.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from MACE (Major Adverse Clinical Events) and/or Device related events during the procedure | during procedure
  MACE defined as: Death, Myocardial Infarction, Stroke, Emergent surgical revascularization of the target vessel, repeat vascularization of the target vessel, bleeding complication requiring transfusion)
Technical success rate | during procedure
  defined as successfully introduction and deployment of the Lokum L-Quest, and/or the Lokum Amplatz, and/or the Slider Hydrophilic Nitinol Guidewire, and/or the Optimus CoCr Stent, and/or the Optimus PFTE covered BE Stent, and/or the AltoSa-XL-PTA, and/or the AltoSa-XL-Gemini Balloon Catheter according to the respective IFU and without device related deficiencies.

SECONDARY OUTCOMES:
For the Optimus CoCr and Optimus-CVS PTFE-covered stent: Freedom from MACE post-procedure, after 6- and 12-months. | Through study completion, an average of 1 year
  MACE defined as: Death, Myocardial Infarction, Stroke, Emergent surgical revascularization of the target vessel, repeat vascularization of the target vessel, bleeding complication requiring transfusion)
For the Optimus CoCr and Optimus-CVS PTFE-covered stent: Freedom from Device-related serious adverse events (SAE's) post-procedure, after 6- and 12-months | Through study completion, an average of 1 year
  Freedom from Device-Related serious adverse events (SAE's)
Freedom from Target Lesion Revascularization post-procedure, at 6- and 12-months | Through study completion, an average of 1 year
  Defined as freedom from a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, Prof. MD., Study Director — Foundation for Cardiovascular Research and Education

IPD SHARING:
Plan to Share IPD: No